CLINICAL TRIAL: NCT01103531
Title: Aerobic Exercise to Improve Outcomes of Treatment for Methamphetamine Dependence
Brief Title: Exercise to Improve Outcomes of Treatment for Methamphetamine Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Richard Rawson, Professor and Associate Director, UCLA Integrated Substance Abuse Programs, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-08-099; 1R01DA027633 (NIH)
Record Dates: First submitted 2010-03-31; First posted 2010-04-14 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Addiction
Keywords: Methamphetamine; Methamphetamine Dependence; Methamphetamine Treatment; Aerobic Exercise; Resistance Exercise; Brain Imaging; D2 and D3 receptor availability
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Group (Experimental): Participants in this group will be scheduled for 24 exercise training sessions over an 8-week period (three times weekly) and will be supervised by a certified exercise physiologist.
  Interventions: Behavioral: Aerobic and Resistance Exercise
- Education Group (Active Comparator): Participants in this group will meet with a counselor who will present and discuss information that includes topics on health and wellness, and lifestyle topics such as healthy eating, meditation, sleep hygiene, and cancer screening.
  Interventions: Behavioral: Educational information about health topics

INTERVENTIONS:
Behavioral: Aerobic and Resistance Exercise — Aerobic and resistance exercise for 24 exercise training sessions over an 8-week period (three times weekly).
  Arms: Exercise Group
Behavioral: Educational information about health topics — A counselor will meet with participants for 24 sessions (3 times/week) over an 8-week period to present and discuss information that includes topics on health and wellness, and lifestyle topics such as healthy eating, meditation, sleep hygiene, and cancer screening.
  Arms: Education Group

SUMMARY:
The purpose of this study is to assess the effects of an aerobic and strength training exercise program (one that increases the need for oxygen and increases muscle) on the treatment outcomes of 150 individuals in treatment for methamphetamine dependence at Cri-Help. The study will determine if a 60-minute exercise program (three times a week) has an effect (good or bad) on the health and drug use of participants as compared to individuals not participating in an exercise program.

DETAILED DESCRIPTION:
Participants were recruited to the study using various methods, including word of mouth and IRB-approved flyers posted throughout the treatment facility. Onsite study staff screened MA-dependent clients in a private study office and reviewed the informed consent protocol. After completion of informed consent procedures, participants entered a1-2week screening phase to determine eligibility, consisting of medical history, physical exam, laboratory studies, and ECG. Eligible clients were taken through study baseline assessments to inform randomization to study conditions, either an exercise intervention or health education control, using a computerized urn randomization program that stratified clients to conditions based on gender (male/female) and severity of baseline MA use (higher vs. lower severity). The cut-off point for determining lower severity MA use versus higher severity use was identified using data from previous clinical outcome studies that show the median number of days of MA use ranges from16 to 20 days at treatment entry. Hence, we defined "lower severity" as using MA for 18 or fewer days in the previous month, and "higher severity" as using for 19 or more days in the past month. The study's data management center (DMC) maintained the urn randomization program and the records that linked participant identification numbers to study condition. Study interventions were conducted onsite while participants were enrolled in usual care at the residential treatment facility; cases of early discharge from the facility resulted in premature termination from the study.

Participants randomized to the exercise condition received a structured exercise program 3 times a week for 8 weeks. Exercise sessions consisted of a 5-min warm-up, 30 min of aerobic activity on a treadmill, followed by 15 min of weight training and a 5-min cool-down/stretching period. Each session was monitored by a staff exercise physiologist who guided one to two participants at a time. Using heart rate monitors, the exercise physiologist worked closely with each individual participant on exercise days to increase treadmill speed/slope to maintain a heart rate between 60% and 85% of maximum for 30 minutes. Once a participant was able to complete two sets of 15 repetitions of any given exercise, weight was incrementally increased.

A data collection protocol occurred at baseline, and also weekly during the 8-week study period, at termination of the study period, and at 1-, 3-, and 6-months post treatment from the residential program (approximately 7-10 days following completion of the intervention period). Participants were compensated $40 per data collection session.

ELIGIBILITY:
Inclusion Criteria:

1. Be seeking treatment for their MA dependence;
2. Be 18 years of age or older, and 45 or younger for males, 55 or younger for females;
3. Meet DSM-IV-TR criteria for MA dependence;
4. Have vital signs that are within clinically acceptable normal range, e.g., resting pulse between 50 and 90 /min, blood pressures between 85-150mm Hg systolic and 45-90mm Hg diastolic;
5. Have a medical history and physical examination that, in the judgment of the study physician or Principal Investigator, show no clinically significant contraindications for study participation;
6. For females, provide negative pregnancy urine tests before randomization (and for the sub-sample, another negative test before the final PET scan at the conclusion of the intervention).

Exclusion Criteria:

1. Clinically significant heart disease or hypertension; unstable pulmonary or cardiovascular disease that would interfere with participation in exercise regimen
2. Neurological or psychiatric disorders as assessed by MINI or clinical interview, such as psychosis, bipolar illness, Tourette's syndrome, major depression, organic brain disease, dementia, or any other neuro-psychiatric disorder that would require ongoing treatment or that would make study compliance difficult;
3. Musculoskeletal disease that would prevent participation in exercise regimen
4. Baseline ECG showing evidence of cardiac ischemia, arrhythmia, or other clinically significant abnormalities
5. Untreated or unstable medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease (other than HIV) that requires immediate medical attention;
6. Clinically significant abnormalities in hematology and chemistry laboratory tests that may make participation hazardous;
7. Have HIV and unable to obtain a clearance for participation from his/her AIDS medical care provider;
8. Pregnant;
9. Any other illness, condition, or use of medications that, in the opinion of the PI and/or the study physician, would preclude safe participation or completion of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2010-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Self-reported Days of Methamphetamine Use | over the 12 week follow-up period
  The primary efficacy measure will be days of self-reported MA use over the 12 weeks after discharge.

SECONDARY OUTCOMES:
Overall Physical Health | 12-week follow-up period
  The effect of the interventions will be compared between the Exercise and Education groups using generalized regression for repeated measures on each of the test results from baseline to discharge to 12 weeks post-discharge
Brain-Imaging Data | End of intervention (9 weeks)
  To examine pre- to post-intervention differences in D2/D3 receptor availability a repeated-measures ANOVA will be performed using the binding potential for [18F]fallypride in subcortical regions of interest.
Psychiatric Symptoms | 12 week follow-up period
  The effect of the interventions will be compared with repeated measures analysis from baseline to discharge to 12 and 26 weeks after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Rawson, PhD, Principal Investigator — UCLA Integrated Substance Abuse Programs
Locations (1):
- Cri-Help, Inc, North Hollywood, California, United States

REFERENCES:
- [Background] Cooper CB. Exercise in chronic pulmonary disease: aerobic exercise prescription. Med Sci Sports Exerc. 2001 Jul;33(7 Suppl):S671-9. doi: 10.1097/00005768-200107001-00005. PMID 11462076
- [Background] Fonkalsrud EW, Mendoza J, Finn PJ, Cooper CB. Recent experience with open repair of pectus excavatum with minimal cartilage resection. Arch Surg. 2006 Aug;141(8):823-9. doi: 10.1001/archsurg.141.8.823. PMID 16927491
- [Background] Glasner-Edwards S, Mooney LJ, Marinelli-Casey P, Hillhouse M, Ang A, Rawson R; Methamphetamine Treatment Project Corporate Authors. Clinical course and outcomes of methamphetamine-dependent adults with psychosis. J Subst Abuse Treat. 2008 Dec;35(4):445-50. doi: 10.1016/j.jsat.2007.12.004. Epub 2008 Feb 21. PMID 18294802
- [Background] Glasner-Edwards S, Mooney LJ, Marinelli-Casey P, Hillhouse M, Ang A, Rawson R; Methamphetamine Treatment Project. Identifying methamphetamine users at risk for major depressive disorder: findings from the methamphetamine treatment project at three-year follow-up. Am J Addict. 2008 Mar-Apr;17(2):99-102. doi: 10.1080/10550490701861110. PMID 18393051
- [Background] Glasner-Edwards S, Mooney LJ, Marinelli-Casey P, Hillhouse M, Ang A, Rawson R; Methamphetamine Treatment Project. Risk factors for suicide attempts in methamphetamine-dependent patients. Am J Addict. 2008 Jan-Feb;17(1):24-7. doi: 10.1080/10550490701756070. PMID 18214719
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1423-34. doi: 10.1249/mss.0b013e3180616b27. PMID 17762377
- [Background] Lautenschlager NT, Cox KL, Flicker L, Foster JK, van Bockxmeer FM, Xiao J, Greenop KR, Almeida OP. Effect of physical activity on cognitive function in older adults at risk for Alzheimer disease: a randomized trial. JAMA. 2008 Sep 3;300(9):1027-37. doi: 10.1001/jama.300.9.1027. PMID 18768414
- [Background] Malek MH, Fonkalsrud EW, Cooper CB. Ventilatory and cardiovascular responses to exercise in patients with pectus excavatum. Chest. 2003 Sep;124(3):870-82. doi: 10.1378/chest.124.3.870. PMID 12970011
- [Background] Monterosso JR, Ainslie G, Xu J, Cordova X, Domier CP, London ED. Frontoparietal cortical activity of methamphetamine-dependent and comparison subjects performing a delay discounting task. Hum Brain Mapp. 2007 May;28(5):383-93. doi: 10.1002/hbm.20281. PMID 16944492
- [Background] Palmer JA, Palmer LK, Michiels K, Thigpen B. Effects of type of exercise on depression in recovering substance abusers. Percept Mot Skills. 1995 Apr;80(2):523-30. doi: 10.2466/pms.1995.80.2.523. PMID 7675585
- [Background] Rawson RA, Anglin MD, Ling W. Will the methamphetamine problem go away? J Addict Dis. 2002;21(1):5-19. doi: 10.1300/j069v21n01_02. PMID 11831500
- [Background] Rawson RA, Marinelli-Casey P, Anglin MD, Dickow A, Frazier Y, Gallagher C, Galloway GP, Herrell J, Huber A, McCann MJ, Obert J, Pennell S, Reiber C, Vandersloot D, Zweben J; Methamphetamine Treatment Project Corporate Authors. A multi-site comparison of psychosocial approaches for the treatment of methamphetamine dependence. Addiction. 2004 Jun;99(6):708-17. doi: 10.1111/j.1360-0443.2004.00707.x. PMID 15139869
- [Background] Simon SL, Domier C, Carnell J, Brethen P, Rawson R, Ling W. Cognitive impairment in individuals currently using methamphetamine. Am J Addict. 2000 Summer;9(3):222-31. doi: 10.1080/10550490050148053. PMID 11000918
- [Background] Simon SL, Domier CP, Sim T, Richardson K, Rawson RA, Ling W. Cognitive performance of current methamphetamine and cocaine abusers. J Addict Dis. 2002;21(1):61-74. doi: 10.1300/j069v21n01_06. PMID 11831501
- [Background] Skrede A, Munkvold H, Watne O, Martinsen EW. [Exercise contacts in the treatment of substance dependence and mental disorders]. Tidsskr Nor Laegeforen. 2006 Aug 10;126(15):1925-7. Norwegian. PMID 16915316
- [Background] Marques-Magallanes JA, Koyal SN, Cooper CB, Kleerup EC, Tashkin DP. Impact of habitual cocaine smoking on the physiologic response to maximum exercise. Chest. 1997 Oct;112(4):1008-16. doi: 10.1378/chest.112.4.1008. PMID 9377910
- [Derived] Salem BA, Gonzales-Castaneda R, Ang A, Rawson RA, Dickerson D, Chudzynski J, Penate J, Dolezal B, Cooper CB, Mooney LJ. Craving among individuals with stimulant use disorder in residential social model-based treatment - Can exercise help? Drug Alcohol Depend. 2022 Feb 1;231:109247. doi: 10.1016/j.drugalcdep.2021.109247. Epub 2021 Dec 31. PMID 34999268
- [Derived] Rawson RA, Chudzynski J, Mooney L, Gonzales R, Ang A, Dickerson D, Penate J, Salem BA, Dolezal B, Cooper CB. Impact of an exercise intervention on methamphetamine use outcomes post-residential treatment care. Drug Alcohol Depend. 2015 Nov 1;156:21-28. doi: 10.1016/j.drugalcdep.2015.08.029. Epub 2015 Sep 3. PMID 26371404
- [Derived] Mooney LJ, Cooper C, London ED, Chudzynski J, Dolezal B, Dickerson D, Brecht ML, Penate J, Rawson RA. Exercise for methamphetamine dependence: rationale, design, and methodology. Contemp Clin Trials. 2014 Jan;37(1):139-47. doi: 10.1016/j.cct.2013.11.010. Epub 2013 Nov 28. PMID 24291456